CLINICAL TRIAL: NCT01784991
Title: "Does a 1 Plus 1 Hydromorphone Pain Protocol Have a Similar Rate of Respiratory Depression to Physician Discretion Protocol in a Geriatric Population With Moderate to Severe Pain?"
Brief Title: Study of Respiratory Depression When Using a Hydromorphone Pain Protocol
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty in recruiting
Sponsor: Albert Einstein Healthcare Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HN - 4325
Record Dates: First submitted 2012-06-25; First posted 2013-02-06 (Estimated); Results first posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2016-12

CONDITIONS: Pain; Respiratory Depression
Keywords: Pain; Opioids; Hydromorphone; regimen
MeSH Terms: conditions — Pain; Respiratory Insufficiency | interventions — Hydromorphone; Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1mg + 1mg Hydromorphone (Active Comparator): Patient will receive 1 mg of hydromorphone for pain at timepoint 0. After 15 minutes, patients will be asked if the still need pain medication. If yes, patients will immediately receive 1mg hydromorphone. Patients will be under continuous monitoring for respiratory depression via capnometer. At 60 minutes, pain will be re-assessed for a second time. If needed, physician will give additional pain meds per their discretion.
  Interventions: Drug: Hydromorphone
- Usual Care Group (Active Comparator): Patient will receive pain medicine per doctor's discretion at timepoint 0. After 15 minutes, patients will be asked if they still need pain medication. If yes, physicians will not be notified and patient will continue to have pain managed as deemed necessary by physician per "usual care." Patients will be under continuous monitoring for respiratory depression via capnometer. At 60 minutes, pain will be re-assessed for a second time. If needed, physician will give additional pain meds per their discretion.
  Interventions: Drug: Usual care group

INTERVENTIONS:
Drug: Hydromorphone — 1mg of Hydromorphone at timepoint 0 and 1 mg of hydromorphone at 15 min timepoint.
  Other Names: Dilaudid
  Arms: 1mg + 1mg Hydromorphone
Drug: Usual care group — Patient will have pain treated at timepoint 0 as per usual care based on physician discretion. At 15 min timepoint, patients will be asked for pain level, and then subsequently treated as per physician discretion.
  Other Names: Morphine; Dilaudid; Other IV opioid medications
  Arms: Usual Care Group

SUMMARY:
This is a study about the efficiency and safety of a 1mg+1mg hydromorphone pain management protocol for the treatment of moderate to sever pain in the Emergency Department. Appropriate patients 60 years and older who present with a condition that causes moderate to severe pain, according to the attending physician's judgment, in which the physician would order the use of parenteral analgesia will be enrolled in one of two study arms, "1+1" versus usual care group. 1+1 patients will receive 1mg hydromorphone followed by another 1mg after 15 minutes if pain persists. Usual care group patients will have pain treated per the discretion of the attending physician. Respiratory status, vital signs, and pain scores will be monitor to assess the efficiency of pain control as well as the safety of pain medicine administration in terms of respiratory depression.

DETAILED DESCRIPTION:
This is a study about the efficiency and safety of a 1mg+1mg hydromorphone pain management protocol for the treatment of long bone fractures in the Emergency Department. Appropriate patients 60 years and older who present with a condition that causes moderate to severe pain, according to the attending physician's judgment, in which the physician would order the use of parenteral analgesia will be screened and randomized to one of two study arms, "1+1" versus usual care group. Neither the research associate, nurse, or attending physician will be blinded to the patients randomization. Patient pain score will be assessed at baseline using VAS score. "1+1" patients will receive 1mg hydromorphone at "timepoint 0" (baseline) followed by another 1mg after 15 minutes (along with repeat VAS pain score) if the patient answers "yes" to "Do you need more pain medicine?" At 60 minutes, patient pain will be assessed a final time and if patient needs more pain medicine, additional treatment will be dictated by physician discretion. Usual care group patients will also have VAS pain scores assessed at timepoint 0, 15 and 60 minutes and will have pain treated per the discretion of the attending physician. Patients will be placed on capnometer for continuous monitoring of respiratory status to guard against any opioid induced respiratory depression. Respiratory status, vital signs, and pain scores will be monitor to assess the efficiency of pain control as well as the safety of pain medicine administration in terms of respiratory depression. We propose that the "1+1" hydromorphone protocol is easy to implement, as it includes a set timeline, a standard question, and a set dosage of a potent analgesic. We hypothesize that it will provide adequate analgesia in the majority of patients without causing the anticipated level of respiratory depression.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient who presents a condition that causes moderate to severe pain, according to the attending physician's judgment, in which the physician would order the use of parenteral analgesia
2. Able to provide consent.

Exclusion Criteria:

1. Patient or family member unable to consent
2. Altered mental status
3. SpO2 less than 95 percent
4. Allergy to opiates
5. Hypotension (Systolic blood pressure less than 90 mmHg)
6. Chronic oxygen dependency or known CO2 retention
7. Acute ETOH or drug intoxication
8. History of chronic pain syndrome or chronic use of opiate narcotics
9. History of opiate/heroin addiction, past or current.
10. End stage renal disease/dialysis patient
11. Chronic metabolic acidosis
12. Physician feels that patient would be poor candidate for study
13. Weight less than 100 pounds, all patients will be weighted
14. Patients younger than 60 years of age

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2014-04-16 (Actual); Study Completion 2014-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Deitch, DO, Principal Investigator — Albert Einstein Medical Center
Locations (1):
- Albert Einstein Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Pre-assignment Details: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Period: Overall Study
Arm/Group | 1mg + 1mg Hydromorphone | Usual Care Group
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Groups:
- Total: Total of all reporting groups
Arm/Group | 1mg + 1mg Hydromorphone | Usual Care Group | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Respiratory Depression
Description: Incidence of respiratory depression (defined as a ETCO2 of 50 mmHg or greater, a 10% change from baseline, or loss of waveform for 15 seconds or greater)
Time Frame: From administration of drug (time 0 minutes) to end of study (60 minute mark)
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | 1mg + 1mg Hydromorphone | Usual Care Group
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Successful Treatment of Patient Pain
Description: Defined as: Declining additional pain medication at 15 minutes or requesting additional pain medication at 15 min, but declining at 60 minutes
Time Frame: 15 min and 60 min after baseline
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | 1mg + 1mg Hydromorphone | Usual Care Group
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in VAS Score
Description: A 13 mm change or greater on a VAS score
Time Frame: 15 min and 60 min after baseline
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | 1mg + 1mg Hydromorphone | Usual Care Group
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Hypoxia
Description: Defined as SpO2 of 93% or less for 15 seconds
Time Frame: From administration of drug (time 0 minutes) to end of study (60 minute mark)
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | 1mg + 1mg Hydromorphone | Usual Care Group
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Hypotension
Description: Hypotension defined as systolic blood pressure less than 90 mmHg
Time Frame: Every 5 minutes from administration of drug (time 0 minutes) to end of study (60 minute mark)
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | 1mg + 1mg Hydromorphone | Usual Care Group
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Allergic Reaction to Study Drug
Time Frame: From administration of drug (time 0 minutes) to end of study (60 minute mark)
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | 1mg + 1mg Hydromorphone | Usual Care Group
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Serious Adverse Events
Description: Defined as prolonged hypoxia, need for positive pressure ventilation or intubation, hospital admission secondary to study drug.
Time Frame: From administration of drug (time 0 minutes) to end of study (60 minute mark)
Population: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | 1mg + 1mg Hydromorphone | Usual Care Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Description: 0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available
Arm/Group | 1mg + 1mg Hydromorphone | Usual Care Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
0 Participants analyzed. PI has left the institution. Efforts made to contact were unsuccessful. No data available

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes